CLINICAL TRIAL: NCT03514355
Title: Pilot Study of Mindfulness-Based Stress Reduction (MBSR) in Patients With Rheumatoid Arthritis That Still Screen Depressed, Despite Adequate Control of Inflammation
Brief Title: MBSR in Rheumatoid Arthritis Patients With Controlled Disease But Persistent Depressive Symptoms
Acronym: PARIS-D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Canadian Initiative for Outcomes in Rheumatology Care (Other)
Responsible Party: Principal Investigator, Gilles Boire, Professor and Rheumatologist, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MP-31-2017-1558
Record Dates: First submitted 2017-08-18; First posted 2018-05-02 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Rheumatoid Arthritis; Depressive Symptoms
MeSH Terms: conditions — Arthritis, Rheumatoid; Depression | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Intervention Model Description: Randomization of consenting eligible patients in intervention and control groups using separate permutated random blocks of 4
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Mindfulness-Based Stress Reduction (MBSR) is a program intended to draw upon the group's shared experiences to facilitate the development of mindfulness. MBSR is offered in 2.5-h classes on a weekly basis for 8 consecutive weeks, with a retreat day in between classes 6 and 7. This day involves guided meditations, allowing for continuity in practice. Classes include specific exercises (e.g. identifying thoughts, emotions and body sensations associated with illness); these are then extended as homework and discussed in the subsequent class. The curriculum themes and content are arranged week by week to reflect these principles.
  Interventions: Behavioral: Mindfulness-Based Stress Reduction
- Control (No Intervention): The control group will receive usual care, with no treatment restrictions. Treating physicians will be informed of CES-D results. Patients will be asked to fulfill the same clinical assessment and questionnaires, and to provide the same biosamples than those patients in the intervention.

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction — 8 weekly 2.5 h sessions plus one day of practice
  Arms: Intervention

SUMMARY:
Despite their efficacy at controlling joint inflammation, current treatments of rheumatoid arthritis (RA) leave up to 40% of patients into non-remission.

Non-remission is most frequently due to persistently negative self-reported global impact of RA, and not to remaining swollen joints or elevated levels of acute phase reactants. In a cohort of recent-onset RA patients diagnosed early and treated to remission (Sherbrooke Early Undifferentiated PolyArthritis (EUPA) cohort), treatment of active disease rapidly led to reduced depressive symptoms in most, but 20% still expressed elevated depressive symptoms (using the CES-D screening tool) after a mean of 7 months. Elevated CES-D scores at this early time strongly predicted never reaching remission over the following 4 years. Elevated CES-D scores were strongly correlated with increased levels of patient-related outcomes (PROs such as fatigue, pain, sleep quality, stiffness and functional limitation), but not with joint or systemic inflammation. In fact, 80% of patients expressing depressive symptoms had controlled joint disease at the same visit. The investigators propose that addressing depressive symptoms will improve RA patients' symptoms and quality of life. In clinical practice, the best indicator of depressive symptoms is the presence of a disconnect between the Patient's (Pt-VAS) and the Physician's (MD-VAS) evaluation of disease activity in patients without objective signs of inflammation.

This pilot study will explore the feasibility and acceptability of testing MBSR in these patients. It will assess over 6 months the changes in depressive symptoms and PROs both in controls and MBSR-treated patients. If positive, the investigators plan to complete a multicenter 6-month Randomized Clinical trial (RCT) (with a 2 year follow up) to formally address the risks/benefits of group MBSR interventions in RA patients with controlled inflammatory disease but positive disconnect between Pt-VAS and MD-VAS.

DETAILED DESCRIPTION:
This is a pilot project for a pragmatic multisite, 6-month, two arm RCT of an MBSR intervention in RA patients expressing depressive symptoms despite controlled joint inflammation, on measures of depressive symptoms (Primary outcome). The investigators will also explore the impact of MBSR on significant PROs (e.g. fatigue, pain, Pt-VAS, anxiety) further translating into lower SDAI scores post-MBSR, and the feasibility of determining if improvement may be mediated though better adherence to treatment and/or through a modification of inflammation-related biomarkers.

During the present 1-year pilot study, the investigators propose to randomize 50 patients, and offer 2 MBSR groups of ≈13 patients each. Due to the bidirectional relationship between RA and depression, MBSR will be studied in patients receiving stable doses of arthritis medications during remission or low disease activity. To avoid recruitment based on thresholds of composite scores (e.g. SDAI) that are strongly impacted by depression-sensitive variables, such as Patient global evaluation of disease activity (PtVAS) and tender joint counts (TJC), the investigators will use a Swollen Joint Count (SJC) ≤2 out of 66 joints and C-Reactive Protein (CRP) ≤8 mg/L ('objective' measures) to define controlled disease. As SJC is the major determinant for RA treatment change in clinical practice, short-term RA treatment changes are unlikely in the recruited patients.

Controlled RA patients reporting Pt-VAS superior to MD-VAS by at least 20/100 units will be recruited. Blinded clinical assessors will determine the joint counts and the Examiner global evaluation of disease activity (EVAS) to determine SDAI scores at baseline and at 6 months. The French Canadian version of the CES-D and the Beck Depression Inventory to assess the importance of depressive symptoms, as well as 0-100 VAS scales (fatigue; sleep; pain; PtVAS) and Health Assessment Questionnaire (HAQ) will be obtained at both visits. Reporting will conform to the CONSORT recommendations for pilot studies.

This study reflects clinical practice, where there is heterogeneity in duration of disease, gender, age, type and dose of RA drugs used, as well as type and dose of antidepressants (when used). While the investigators suggest that RA drugs remain constant over the 6-month intervention period, treating physicians will be free to modify treatment if clinically indicated. Antidepressant use will not be an exclusion criterion.

For pragmatic reasons (e.g. uneven availability and expertise of primary care physician's (PCP), unknown effect size of the intervention), the investigators will not include a second active treatment arm with optimization of antidepressants. Instead, the investigators will inform in writing treating PCPs of their patient participation to the study and of the disconnect between Pt-VAS and MD-VAS. Changes to arthritis and depression drugs will be tracked and controlled for in analyses. For patients' safety, psychological contraindications to MBSR will be screened at baseline during a phone interview by Dr Françoise Gendron who will direct the MBSR sessions, and patients with contraindications excluded.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years, with stable (3 months) disease modifying antirheumatic drugs (DMARDs) and/or biologic-treated RA (meeting classification criteria)
2. both ≤2/66 SJC plus CRP ≤8 mg/L
3. Patient Evaluation of disease activity (Pt-VAS) ≥20 higher than Physician Evaluation of Disease Activity (MD-VAS).

Exclusion Criteria:

1. Inability to consent (e.g. not fluent in French, dementia) or to participate in groups;
2. Active vasculitis, SJC ≥3, CRP ≥8, arthritis drug changes (i.e. addition or increase of DMARDs or biologics or oral corticosteroids) during the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2017-09-04 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2021-09-29 (Actual)

PRIMARY OUTCOMES:
Spontaneous variation in Center for Evaluation Studies - Depression (CES-D) score in controls | 6 months
  to estimate the variations in CES-D scores (range 0-60; depression suggested if at least 16) between baseline and 6 months (i.e. about 3 months after the end of MBSR) in the randomized controls

SECONDARY OUTCOMES:
Numbers of patients recruited using current recruitment strategy | 6 months
  adjust recruitment strategy to obtain an optimal one, that is being able to form randomized groups of 15 patients in the MBSR group and 15 controls, every 6 months over 12 months
Impact of Mindfulness-Based Stress Reduction (MBSR) on Patient evaluation of disease activity of Rheumatoid arthritis | 6 months
  to estimate the impact of MBSR on Patient evaluation of disease activity of Rheumatoid arthritis (range 0-10, 0 meaning no disease activity and 10 the most active disease possible according to the patient) between baseline and 6 months following MBSR
Impact of Mindfulness-Based Stress Reduction (MBSR) on Center for Epidemiologic Studies Depression Scale Revised (CES-D) depressive symptoms) | 6 months
  to estimate the impact of MBSR on Center for Epidemiologic Studies Depression Scale Revised between baseline and 6 months following MBSR. The scale goes from 0 to 60 (60 meaning the maximal depressive symptoms possible). An individual from the general population with a score above 16 is considered with possible depression and a clinical assessment for depression may be justified; the equivalent threshold in patients with rheumatoid arthritis is 19.
Impact of MBSR on anxiety | 6 months
  estimate impact of MBSR (versus control) between baseline and 6 months on anxiety measured using the Generalized Anxiety Disorder-7 (GAD-7 scale from 0 to 21, 21 being the worst possible score)
Impact of MBSR on pain | 6 months
  estimate impact of MBSR (versus control) between baseline and 6 months on pain (Visual Analog Scale goes from 0-100, with 100 indicating the most severe possible pain)
Impact of MBSR on fatigue | 6 months
  estimate impact of MBSR (versus control) between baseline and 6 months on fatigue (Visual Analog Scale goes from 0 to100, with 100 indicating the most severe fatigue possible)
Beck Depression Inventory (BDI) | 6 months
  Impact of MBSR (versus control) between baseline and 6 months on BDI scores (range 0-63, 63 being the worst possible score)
Numbers of patients with complete Biomarker collection | 6 months
  validate our methods of biomarker collection to attain more than 90% of usable samples
Numbers of patients with adverse events linked to MBSR | 6 months
  track adverse events associated with MBSR in RA patients according to CTCAE v4.03

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Boire, MD, MSc, Principal Investigator — Université de Sherbrooke
Locations (1):
- Centre intégré universitaire de santé et de services sociaux (CIUSSS) de l'Estrie - CHUS, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No